CLINICAL TRIAL: NCT00054951
Title: A Phase I/II, Open Label, Multicenter, Single-Arm, Safety and Efficacy Study of Doxorubicin Hydrochloride Adsorbed to Magnetic Targeted Carriers (MTC-DOX) Administered by Intrahepatic Delivery (Via Hepatic Artery Catheterization) for the Treatment of Patients With Unresectable Hepatocellular Carcinoma.
Brief Title: Safety and Efficacy of Doxorubicin Adsorbed to Magnetic Beads
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: FeRx (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTC-DOX-006
Record Dates: First submitted 2003-02-13; First posted 2003-02-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatoma; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Injections

INTERVENTIONS:
Drug: MTC-DOX for Injection

SUMMARY:
MTC-DOX is Doxorubicin or DOX, a chemotherapy drug, that is adsorbed, or made to "stick," to magnetic beads (MTCs). MTCs are tiny, microscopic particles of iron and carbon. When DOX is added to MTCs, DOX attaches to the carbon part of the MTCs. MTC-DOX is directed to and deposited in the area of a tumor, where it is thought that it then "leaks" through the blood vessel walls. Once in the surrounding tissues, it is thought that Doxorubicin becomes "free from" the magnetic beads and will then be able to act against the tumor cells. The iron component of the particle has magnetic properties making it possible to direct MTC-DOX to specific tumor sites in the liver by placing a magnet on the body surface. It is hoped that MTC-DOX used with the magnet may target the chemotherapy directly to liver tumors and provide a treatment to patients with liver cancer.

Patients enrolled in the study will be administered MTC-DOX through a hepatic artery catheter inserted under radiological guidance. During and following injection of the MTC-DOX, the drug will be localized to the hepatic tumor site by use of an external magnet. Dose may be divided in order to localize MTC-DOX to all lesions. The MTC-DOX intrahepatic infusions will be repeated every three weeks until tumor progression, complete remission, unacceptable toxicity, or a maximum of six treatment cycles.

The purpose of this Phase 1/2 study is to evaluate time to disease progression following administration of MTC-DOX.

ELIGIBILITY:
Patients may be enrolled into this protocol only if all of the following inclusion criteria are met:

* Patient has unresectable hepatocellular carcinoma diagnosed by CT scan and meets criteria described in Section 23.
* Total combined cross-sectional area of all hepatic tumors as determined by CT scan is between 4 and 150 cm2.
* The center of the tumor(s) mass must be less than or equal to 14 cm from the anterior lateral abdominal wall as determined by cross-sectional imaging at baseline. This is required for optimal placement of the magnet. If more than one tumor mass is present, all of the tumor masses must meet this criterion.
* Patient is ambulatory with a Karnofsky performance status score greater than or equal to 60 and an estimated life expectancy of greater than or equal to 3 months.
* Patient is between 18 and 80 years old.
* Patient is judged by the investigator to have the initiative and means to be compliant with the protocol and be within geographical proximity to allow follow-up.
* Patient or legal representative has the ability to give informed written consent prior to initiation of therapy.
* If patient is female and of childbearing potential, she must have a negative b-HCG prior to receiving treatment.
* Patient must agree to use an effective method of contraception (e.g., birth control pills, condoms, intrauterine device, diaphragm, Norplant, Depo-Provera).

Patients will be excluded from enrollment if any of the following apply:

* Patient has a history of cancer other than hepatocellular (excluding resected basal cell carcinoma; or curatively resected stage 1 or less cervical cancer if disease free for 5 years or more).
* Patient has had prior radiation therapy within the last 6 months or chemotherapy within the last 4 weeks.
* Patients with diffuse hepatocellular carcinoma or disease that precludes delivery of the drug to the tumor via a vessel that feeds the tumor.
* Patient has another active medical condition(s) or organ disease(s) that may either compromise patient safety or interfere with the safety and/or outcome (e.g., survival) evaluation of the study drugs. While this exclusion is not limited to the following abnormalities, if any of the following laboratory abnormalities are present, the patient should be excluded:

WBC < 3,500/uL Platelets < 40,000/ul Hemoglobin < 9.5 gm/dL Total bilirubin > 2.5 mg/dL ALT or AST > or equal to 5 x upper limit of normal Serum Creatinine > 2.0 mg/dL INR > or equal to 2.0

* Patient has cardiac dysfunction with a left ventricular ejection fraction < 40%.
* Patient or physician plans concomitant chemotherapy, radiation therapy, hormonal and/or biological treatment for cancer including immunotherapy (excluding megace, oral contraceptives or post menopausal estrogen replacement therapy) while on study.
* Patients with an indwelling cardiac pacemaker, cerebral aneurysm clips, or any other indwelling device or appliance that could be adversely affected by the use of the external magnet.
* Patients with documented evidence of hemachromatosis or hemosiderosis.
* Patients with CT or Ultrasound evidence of main or first branch portal vein invasion or thrombosis.
* Prior orthotopic hepatic transplant.
* Patient has received previous treatment with doxorubicin, idarubicin, and/or other anthracyclines or anthracenes.
* Patient has a known allergy to doxorubicin, MTC-DOX or any of their components.
* Patient has been treated with any investigational drug, investigational biologic, or investigational therapeutic device within 30 days of initiating study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: Joy Koda, Ph. D., Study Director — VP Clinical Development
Locations (3):
- China (3):
  - Cancer Institute & Hosp. CAMS, Beijing
  - Chinese PLA Cancer Ctr. Yang Gongjing, Nanjing
  - Zhong Shan Hospital, Fudan University, Shanghai